CLINICAL TRIAL: NCT03696784
Title: A Phase I Study of Autologous Activated T-cells Targeting the CD19 Antigen and Containing the Inducible Caspase 9 Safety Switch in Subjects With Relapsed/Refractory B-cell Lymphoma
Brief Title: Anti-CD19 CAR-T Cells With Inducible Caspase 9 Safety Switch for B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: UNC Chapel Hill University Cancer Research Fund (Unknown); The V Foundation (Other); M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1813-ATL; K12CA120780 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases
Keywords: CAR T cells; CD19; Lymphoma; AP1903; Cytokine Release Syndrome; Neurotoxicity; Rimiducid
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Cytokine Release Syndrome; Neurotoxicity Syndromes | interventions — Bendamustine Hydrochloride; fludarabine; fludarabine phosphate; AP 1903 reagent; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Arm iC9.CAR19 T cells (Experimental): The safety of iC9-CAR19 cells will be investigated using the 3+3 design. Dose level (DL) Dose (#transduced cells/kg)
  -1 1 x 10^5
  1. 1 x 10^6
  2. 2 x 10^6 DL1 will enroll 3 subjects. If no toxicity within 4 weeks, then DL 2 will enroll 3 subjects. If toxicity in 1/3 subjects in DL 1, 3 more subjects will be enrolled. If DL 1 is not tolerable, a de-escalation to DL -1 will enroll 3 subjects. If 3 subjects at the higher dose do not have DLTs more will be enrolled at that dose to get more information about toxicity.
  Lymphodepleting chemotherapy of IV bendamustine 70 mg/m2 and IV fludarabine 30 mg/m2/day for 3 consecutive days will be given within 2-14 days prior to cell infusion.
  AP1903 (0.4 mg/kg), a dimerizing agent to engage and activate the caspase 9 safety switch to trigger iC9-CAR19 T cell death by apoptosis will be given to subjects who develop severe cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS).
  Interventions: Biological: iC9-CAR19 T cells; Drug: Bendamustine; Drug: Fludarabine; Drug: AP1903; Drug: Cyclophosphamide
- Expansion Cohort iC9-CAR19 cells (Experimental): After the tolerable cell dose (TCD) has been determined in adults, up to 18 additional subjects may be enrolled in an expansion cohort at the TCD. A TCD is defined as the dose at which approximately 0.20 of subjects experience dose limiting toxicity (0 - 1 out of 6 subjects).
  Interventions: Biological: iC9-CAR19 T cells; Drug: Bendamustine; Drug: Fludarabine; Drug: AP1903; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: iC9-CAR19 T cells — iC9-CAR19 T cells will be given by a licensed healthcare provider via intravenous injection over 5-10 minutes through either a peripheral or a central line.
Drug: Bendamustine — 70mg/m2 IV given as a daily infusion for 3 days per institutional guidelines 2 - 14 days prior to the T cell infusion.
  Other Names: Treanda; Bendeka
Drug: Fludarabine — 30 mg/m2 given as a daily infusion for 3 days per institutional guidelines 2 - 14 days prior to the T cell infusion
  Other Names: Fludara
Drug: AP1903 — 0.4 mg/kg of AP1903 as an IV infusion over 2 hrs for subjects who develop Grade 4 cytokine release syndrome (CRS) or grade ≥3 CRS that is unresponsive to standard of care interventions , subjects who develop grade ≥3 Immune effector cell-associated neurotoxicity syndrome (ICANS) that does not improve to grade ≤1 within 72 hours with standard of care interventions, and subjects with grade 4 ICANS of any duration that have evidence of cerebral edema and/or generalized convulsive status epilepticus.
  Subjects in the expansion cohort who experience ≥ grade 2 CRS or ICANS that remains ≥ grade 2, twenty-four hours after an initial dose of the standard of care treatment may be part of the sub-study of rimiducid. These subjects will receive one of two assigned dose levels. DL1 and DL2 doses are 0.05 mg/kg and 0.01 mg/kg for subjects and DL1: 0.1 mg/kg and DL2: 0.01 mg/kg for subjects with ICANS.
  Other Names: Rimiducid
Drug: Cyclophosphamide — 500 mg/m2/day administered by IV over 3 consecutive days
  Other Names: Cytoxan; Neosar

SUMMARY:
This research study combines 2 different ways of fighting disease: antibodies and T cells. Both antibodies and T cells have been used to treat patients with cancers, and both have shown promise, but neither alone has been sufficient to cure most patients. This study combines both T cells and antibodies to create a more effective treatment. The treatment being researched is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD19 antigen (ATLCAR.CD19) administration.

Prior studies have shown that a new gene can be put into T cells and will increase their ability to recognize and kill cancer cells. The new gene that is put in the T cells in this study makes a piece of an antibody called anti-CD19. This antibody sticks to leukemia cells because they have a substance on the outside of the cells called CD19. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood part of it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD19 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

Preliminary results have shown that subjects receiving this treatment have experienced unwanted side effects including cytokine release syndrome and neurotoxicity. In this study, to help reduce cytokine release syndrome and/or neurotoxicity symptoms, the ATLCAR.CD19 cells have a safety switch that, when active, can cause the cells to become dormant. These modified ATLCAR.CD19 cells with the safety switch are referred to as iC9-CAR19 cells. If the subject experiences moderate to severe cytokine release syndrome and or neurotoxicity as a result of being given iC9-CAR19 cells, the subject can be given a dose of a second study drug, AP1903, if standard interventions fail to alleviate the symptoms of cytokine release syndrome and/or neurotoxicity. AP1903 activates the iC9-CAR19 safety switch, reducing the number of the iC9-CAR19 cells in the blood. The ultimate goal is to determine what dose of AP1903 can be given that reduces the severity of the cytokine release syndrome and/or neurotoxicity, but still allows the remaining iC9-CAR19 cells to effectively fight the lymphoma.

The primary purpose of this study is to determine whether receiving iC9-CAR19 cells is safe and tolerable in patients with relapsed/refractory B-cell lymphoma, primary central nervous system lymphoma and chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
This study is a phase I dose finding trial to determine if chimeric antigen receptor T (CAR-T) cells targeting the CD19 antigen and containing the inducible caspase 9 safety switch can be safely administered to adult subjects with relapsed or refractory B-cell Lymphoma, primary central nervous system lymphoma and chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL). The safety of iC9-CAR19 cells will be investigated using the 3+3 design. The starting dose of 1 x 106 transduced cells/kg (dose level 1) will enroll at least 3 subjects in the initial cohort. If there are no dose limiting toxicities (DLTs) within 4 weeks of the cell infusion in these 3 subjects, then the next cohort will evaluate 2 x 106 transduced cells/kg. If there is toxicity in 1/3 subjects in the initial cohort, the cohort will be expanded to enroll up to 6 subjects. During iC9-CAR19 T cell dose exploration, rimiducid (0.4 mg/kg), a dimerizing agent that is designed to engage and activate the caspase 9 safety switch to trigger iC9-CAR19 T cell death by apoptosis will be given to subjects who develop grade 4 cytokine release syndrome (CRS) or grade ≥3 CRS that is unresponsive to standard of care interventions, and to subjects who develop grade ≥3 Immune effector cell-associated neurotoxicity syndrome ( ICANS) that does not improve to grade ≤1 within 72 hours with standard of care interventions, and subjects with grade 4 ICANS of any duration that have evidence of cerebral edema and/or generalized convulsive status epilepticus. After the tolerable cell dose (TCD) of iC9-CAR19 T cells has been determined, up to 18 additional adult subjects may be enrolled in an expansion cohort at the TCD. Rimiducid will be given to subjects in the expansion cohort who develop grade ≥3 immune effector cell-associated neurotoxicity syndrome (ICANS) that does not improve to grade ≤1 within 72 hours with standard of care interventions, and subjects with grade 4 ICANS of any duration that have evidence of cerebral edema and/or generalized convulsive status epilepticus. Subjects in the expansion cohort who experience ≥grade 2 CRS or ICANS that remains ≥grade 2 twenty-four hours after initial standard of care treatment (tocilizumab for CRS or steroids for ICANS) may be part of the rimiducid sub-study. These subjects will receive one of two assigned dose levels of rimiducid with their second standard of care treatment. The percent reduction in CAR T cells will be measured in these subjects. If the subjects' CRS or ICANS is unresponsive to standard treatment and the assigned dose level of rimiducid, subjects with ≥grade3 CRS or ICANS will then be given a full dose (0.4 mg/kg) of rimiducid. If the subject's CRS or ICANS is at grade 2 48 hours after the first dose of rimiducid, they will receive another dose of rimiducid at the assigned dose level.

Cell Procurement Peripheral blood, up to 300 mL (in up to 3 collections) will be obtained from subjects for cell procurement. In subjects with inadequate lymphocyte count in the peripheral blood, a leukapheresis may be performed to isolate sufficient T cells. The parameters for apheresis will be up to 2 blood volumes.

Lymphodepleting Regimen Subjects will receive a "pre-conditioning" cytoreductive regimen of bendamustine 70 mg/m2/day administered IV followed by an IV dose of fludarabine 30 mg/m2/day administered over 3 consecutive days. These agents will be administered per institutional guidelines. Prophylaxis (e.g., hydration, antiemetics, etc.) needed prior to fludarabine and bendamustine chemotherapy will be provided per institutional guidelines. At the discretion of the clinical investigator, subjects with a known history of intolerance to bendamustine may be considered for lymphodepletion with cyclophosphamide 500 mg/m2/day administered by IV followed by an IV dose of fludarabine 30 mg/m2/day administered over 3 consecutive days. These agents will be administered per institutional guidelines.

Administration of iC9-CAR19 T cells Post lymphodepletion, subjects who meet eligibility criteria for cellular therapy will receive iC9-CAR19 T cells within 2 - 14 days after completing the lymphodepleting chemotherapy regimen. Post lymphodepletion iC9-CAR19 will be administered at dose levels specified in the protocol. A recently published trial in refractory DLBCL established that a dose of 2 x 10 6 CAR19+ T cells/kg was safe and associated with significant in vivo expansion and we anticipate similar results with iC9-CAR19+ T cells.

Duration of Therapy Therapy in this study involves 1 infusion of iC9-CAR19 cells.

Duration of Follow-up Subjects who receive a cell infusion will be followed for up to 15 years for replication-competent retrovirus evaluation or until death, whichever occurs first. Subjects who are removed from study and do not receive the cellular therapy product due to unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria for the Study:

Unless otherwise noted, subjects must meet all of the following criteria to participate in all stages of this study:

* Written informed consent and HIPAA authorization for release of personal health information.
* Adults ≥18 years of age.
* Histologically confirmed B-cell NHL, including the following types defined by WHO 2016:

Aggressive Lymphomas:

* DLBCL not otherwise specified (NOS)
* T cell/histiocyte rich large B cell lymphoma; primary cutaneous DLBCL, leg type; EBV-positive DLBCL NOS; DLBCL associated with chronic inflammation; Large B-cell lymphoma with IRF4 rearrangement; Intravascular large B-cell lymphoma; ALK-positive large B-cell lymphoma
* Primary mediastinal (thymic) large B-cell lymphoma
* High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement; high grade B-cell lymphoma, NOS
* B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
* Transformation of indolent lymphoma or CLL to DLBCL will also be included
* Burkitt lymphoma
* Primary CNS lymphoma

Indolent Lymphomas:

* Follicular lymphoma
* Splenic marginal zone lymphoma
* Extranodal marginal zone lymphoma of mucosa-associated lymphoid tissue
* Nodal marginal zone lymphoma
* Waldenstrom's macroglobulinemia (Lymphoplasmacytic lymphoma)
* Mantle cell lymphoma
* CLL/SLL by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria
* Subjects with CNS involvement of lymphoma are eligible.

  --For aggressive lymphomas, must have relapsed or refractory disease after having received at least 2 prior lines of systemic therapy, including, at a minimum:
  * An anti-CD20 monoclonal antibody
  * An anthracycline containing chemotherapy regimen (if eligible)
  * An autologous stem cell transplant (if eligible)
* Subjects with primary CNS lymphoma must have failed at least 1 prior line of therapy that included high dose methotrexate.
* For indolent lymphomas, subjects must have received at least 2 prior lines of therapy for their lymphoma
* Subjects with specifically relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma must have received at least 2 prior therapy regimens which can include, but not limited to:

  * A combination of an anti-CD20 monoclonal antibody and an alkylating agent, OR
  * A Bruton's Tyrosine Kinase Inhibitor, OR
* A BCL-2 inhibitor in combination with an anti-CD20 monoclonal antibody.
* Subjects with prior or concurrent malignancies of the same or different tumor type whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational drug are eligible for enrollment at the discretion of the clinical investigator.
* Subjects relapsed after allogeneic stem cell transplant will be eligible if they meet other inclusion criteria and have no active graft vs host disease (GVHD)
* Measurable or assessable disease by Lugano criteria, response criteria for primary CNS lymphoma, or WM criteria, or IWCLL criteria. Subjects with bone marrow-only involvement are eligible.
* Karnofsky score of > 60%
* Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. WOCBP subjects will also be instructed to tell their male partners to use a condom.

Exclusion Criteria for the Study:

Subjects meeting any of the following exclusion criteria will not be able to participate in this study (procurement, lymphodepletion, and cell infusion):

* Subject is pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Current use of systemic corticosteroids at doses ≥10mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at the discretion of investigator. Patients with primary CNS lymphoma can receive higher doses of steroids per the investigator's discretion.
* Active infection with HIV, HTLV, HBV, and HCV (can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells) defined as not being well controlled on therapy. Subjects are required to have negative HIV antibody, negative HTLV1 and HTLV2 antibodies, negative Hepatitis B surface antigen, and negative HCV antibody or viral load. In addition, subjects with positive Hepatitis B core antibody will have Hepatitis B viral load tested and subjects with positive Hepatitis B viral load will also be excluded.
* Subject must either have core antibody negative HBV (results can be pending at the time of cell procurement) OR if a subject is hepatitis B core antibody positive they must have their hepatitis B viral load checked. These subjects will be excluded if their viral load is positive at baseline. Subjects who are core antibody positive and viral load negative at baseline will be considered eligible.
* A history of intolerance to fludarabine. Note: subjects with history of intolerance to bendamustine may be considered for enrollment at the discretion of the clinical investigator if they are candidates for lymphodepletion with cyclophosphamide and fludarabine.

Eligibility criteria to be met prior to procurement:

* Subjects must sign a consent to undergo cell procurement.
* Life expectancy ≥ 12 weeks.
* Evidence of adequate organ function as defined by:

The following is required within 7 days prior to procurement:

* Bilirubin ≤1.5 times the upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5× ULN)
* AST ≤ 3 times ULN
* Creatinine Clearance (CrCl) >30mL/min per Cockcroft and Gault
* Pulse oximetry of >90% on room air

  * Left ventricular ejection fraction (LVEF) ≥35% as measured by ECHO, with no additional evidence of decompensated heart failure.
  * In patients with disease assessed by imaging, imaging results from within 90 days prior to procurement to assess the presence of active disease. If disease is not measurable by imaging, evidence of active disease within 90 days of procurement via bone marrow biopsy or SPEP/immunofixation.
  * Negative serum pregnancy test within 72 hours prior to procurement or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for >1 year, or documentation of surgical menopause involving bilateral oophorectomy.

Eligibility criteria to be met prior to lymphodepletion:

* Written informed consent to enroll in the CAR T-cell therapy trial must be obtained prior to lymphodepletion.
* Imaging results from within 7 days prior to lymphodepletion. Imaging must occur at least 3 weeks after most recent therapy (used as baseline measure for documentation of progression before the lymphodepletion) to document measurable or assessable disease. Imaging does not need to be repeated if it is within 7 days prior to lymphodepletion. For WM, imaging does not need to be repeated prior to lymphodepletion if no evidence of disease at screening.
* Evidence of adequate organ function as defined by:

The following are required within 72 hours prior to lymphodepletion:

* Adequate bone marrow function (ANC ≥1.0 x 10^9/L and platelets ≥50 x 10^9/L) unless related to lymphoma involvement. Subjects cannot have received platelet transfusion within 7 days of lymphodepletion.
* Bilirubin ≤1.5 times the upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5× ULN)
* AST ≤ 3 times ULN
* Creatinine Clearance (CrCl) >30mL/min per Cockcroft and Gault
* Pulse oximetry of > 90% on room air
* Negative serum pregnancy test within 72 hours prior to lymphodepletion or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for > 1 year, or documentation of surgical menopause involving bilateral oophorectomy.
* In subjects with CLL/SLL or lymphoma with bone marrow only involvement, a bone marrow biopsy within 28 days prior to lymphodepletion.
* Subjects that have received therapy with murine antibodies must have documentation of absence of human anti-mouse antibodies (HAMA) prior to lymphodepletion. Subjects who have received prior therapy with murine antibodies must have documentation of absence of HAMA within 8 weeks of lymphodepletion or after their most recent murine antibody therapy (whichever is shortest). For subjects that receive murine monoclonal antibodies or murine-human chimeric monoclonal antibodies between procurement and lymphodepletion, HAMA testing should be performed within 4 weeks prior to lymphodepletion and after the last monoclonal antibody dose.
* Available autologous transduced activated T cells product meets the certificate of analysis.
* Has not received any investigational agents or received any tumor vaccines within the previous six weeks prior to lymphodepletion.
* Subject is not taking a prohibited or contraindicated medication prior to lymphodepletion. Contraindicated medications should be discontinued at least two weeks prior to the scheduled lymphodepletion or by at least 5 half-lives of the contraindicated medication, whichever is shorter.
* Subject is not taking strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. (This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine).
* Subject has not received chemotherapy within the previous 3 weeks prior to lymphodepletion.

Eligibility criteria to be met prior to cell infusion after lymphodepletion:

* No evidence of uncontrolled infection or sepsis.
* Negative serum pregnancy within 7 days of cell infusion (does not need to be repeated if pre-lymphodepletion pregnancy test is within window).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2040-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of iC9-CAR19 T cells | 4 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. ICANS symptoms will be graded per ASBMT ICANS Consensus Grading for Adults (scale from 1-mild to 4-critical) and cytokine release syndrome (CRS) symptoms will be graded according to ASBMT CRS Consensus Grading (a scale from 1-mild to 5-death).

SECONDARY OUTCOMES:
Identify a recommended phase 2 dose (RP2D) of iC9-CAR19 T cells in subjects with relapsed or refractory B-cell lymphoma or CLL/SLL | 4 weeks
  The recommended phase 2 dose of iC9-CAR19 cells will be determined based on 3+3 dose finding rules and the tolerability of iC9-CAR19 cells assessed by NCI-CTCAE criteria, CRS grading criteria, and ICANS grading criteria.
Survival of iC9-CAR19 T cells in vivo | 15 years
  Persistence of iC9-CAR19 T cells in vivo will be determined by quantitative polymerase chain reaction (PCR) and flow cytometry in samples of peripheral blood.
Overall response rate (ORR) (rate of Complete Response (CR)) mediated by autologous iC9-CAR19 T cells administered to subjects with relapsed or refractory B-cell lymphoma or CLL/SLL | 15 years
  ORR:
  * Revised Lugano criteria CR= no new lesions; normal bone marrow (BM); Target nodes/masses ≤ 1.5 cm; no extra lymphatic sites; and/or PET-CT score of 1-3.
  * For Primary CNS Lymphoma CR= No contrast enhancement on brain imaging; no corticosteroid dose; normal eye exam; negative cerebrospinal fluid (CSF) cytology.
  * For Waldenström Macroglobulinemia (WM) CR= normal Immunoglobulin M (IgM)); no monoclonal protein by immunofixation; no histological evidence of BM involvement; resolution of any adenopathy/organomegaly; no signs or symptoms of WM.
  * International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Revised Criteria Assessment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) CR=Target nodes/nodal masses ≤ 1.5 cm; normal lymphocyte count; platelets > 100E9/L; Hemoglobin > 11.0 g/dL; ANC > 1.5E9/L; no evidence for typical CLL lymphocytes and without nodular lymphoid aggregates on BM biopsy; no constitutional symptoms from CLL/SLL; no hepatosplenomegaly
Overall survival (OS) in subjects with relapsed or refractory B-cell lymphoma or CLL/SLL following infusion of iC9-CAR19 T cells | 15 years
  OS will be measured from the date of administration of iC9-CAR19 T cells to the date of death. Subjects who have not died by the analysis data cut-off date will be censored at their last date of contact.
Progression free survival (PFS) in subjects with relapsed or refractory B-cell lymphoma or CLL/SLL following infusion of iC9-CAR19 T cells | 15 years
  PFS is day of infusion to date of disease progression (PD) or death due to any cause.
  * Lugano criteria PD= PET-CT score 4 or 5 with increase in intensity of uptake from baseline and/or New FDG-avid foci consistent with lymphoma
  * Response Criteria for Primary CNS Lymphoma PD=25% increase in lesion or new site of disease on brain imaging; recurrent/new ocular disease; recurrent/positive CSF cytology
  * Response Criteria for WM PD= ≥ 25% increase in serum IgM or progression of clinically significant findings due to disease; or symptoms attributable to WM
  * IWCLL Revised Criteria for Response Assessment of CLL/SLL PD= New enlarged lymph node > 1.5 cm; new hepato- and/or splenomegaly or organ infiltration; 50% increase from baseline of previous site; 50% increase from baseline of circulating lymphocyte count or CLL cells on marrow biopsy; 50% decrease in platelet count from baseline prior to therapy; Or > 2 gm g/dL decrease in hemoglobin from baseline
Duration of response (DOR) in subjects with relapsed or refractory B-cell lymphoma or CLL/SLL who experience an objective response following infusion of iC9-CAR19 T cells | 15 years
  DOR is defined for subjects who experience an objective response as the date of first objective response to the date of disease progression (per the Lugano criteria, Response Criteria for Primary CNS Lymphoma Response Criteria for WM or IWCLL Revised Criteria for Response Assessment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma) or death as a result of any cause. Subjects who do not meet criteria for progression or death by the analysis cut-off date will be censored at their last evaluable disease assessment date.
Change in patient-reported symptoms | 1 year
  Patient reported symptoms will be measured using selected symptoms from the NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE). The PRO-CTCAE is a patient-reported outcome measurement system developed to characterize the frequency, severity and interference of symptomatic treatment toxicities. Each of the symptom terms included in the PRO-CTCAE is assessed relative to one or more distinct attributes, including presence/absence, frequency, severity, and/or interference with usual or daily activities. Responses are provided on a 5-point Likert scale: Frequency item: How OFTEN did you have? (Never / Rarely / Occasionally / Frequently / Almost constantly); Severity item: What was the SEVERITY of your at its WORST? (None / Mild / Moderate / Severe / Very severe);Interference item: How much did INTERFERE with your usual or daily activities? (Not at all / A little bit / Somewhat / Quite a bit / Very much)
Change in physical function | 1 year
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a v1.0. assesses one's ability to carry out activities that require physical actions, ranging from self-care (activities of daily living) to more complex activities that require a combination of skills, often within a social context. "Physical Function" is inclusive of the term "disability" and includes the full spectrum of physical functioning from severe impairment to exceptional physical abilities. Each question has five response options ranging in value from one to five, resulting in a total score (T-score) from 0 to 100. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Physical Function, a T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
Change in health related quality of life | 1 year
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health measures assess an individual's physical, mental, and social health. The measures are generic, rather than disease-specific, and often use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. Each question has five response options ranging in value from one to five, which are summed into T-score values for physical and mental health. A higher PROMIS T-score represents more of the concept being measured. Thus, a person who has T- scores of 60 for the Global Physical Health or Global Mental Health scales is one standard deviation better (more healthy) than the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/patientcare/clinical-trials